CLINICAL TRIAL: NCT02299414
Title: A Pragmatic Multicenter Randomized Clinical Trial (RCT) of Antihypertensive Therapy for Mild Chronic Hypertension During Pregnancy: Chronic Hypertension and Pregnancy (CHAP) Project
Brief Title: Chronic Hypertension and Pregnancy (CHAP) Project
Acronym: CHAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Columbia University (Other); Drexel University College of Medicine (Other); Rutgers, The State University of New Jersey (Other); Lehigh Valley Hospital (Other); Saint Peters University Hospital (Other); Christiana Care Health Services (Other); Washington University School of Medicine (Other); Duke University (Other); University of Texas Southwestern Medical Center (Other); The University of Texas Health Science Center, Houston (Other); Stanford University (Other); University of Pennsylvania (Other); The University of Texas Medical Branch, Galveston (Other); University of Utah (Other); Intermountain Health Care, Inc. (Other); University of California, San Francisco (Other); Johns Hopkins University (Other); University of Pittsburgh (Other); Ochsner Health System (Other); University of North Carolina, Chapel Hill (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); WakeMed Health and Hospitals (Other); San Francisco General Hospital (Other); McKay-Dee Hospital (Other); Winthrop University Hospital (Other); New York Hospital Queens (Other); Latter Day Saints Hospital (Other); Lyndon B Johnson General Hospital (Other); Virtua Medical Group (Other); Duke Regional Hospital (Other); Utah Valley Regional Medical Center (Other); Northwestern University (Other); Women and Infants Hospital of Rhode Island (Other); Baylor College of Medicine (Other); Case Western/Metro Health (Unknown); Ohio State University (Other); University of Iowa (Other); University of California, San Diego (Other); Indiana University (Other); Meriter Foundation (Other); Weill Medical College of Cornell University (Other); University of Oklahoma (Other); Medical University of South Carolina (Other); Beaumont Hospital (Other); University of Colorado, Denver (Other); University of Kansas Medical Center (Other); Denver Health and Hospital Authority (Other); Gundersen Health System (Other); Wake Forest University Health Sciences (Other); Oregon Health and Science University (Other); Medical College of Wisconsin (Other); Temple University (Other); New Jersey Medical School (Other); University of South Alabama (Other); Vanderbilt University (Other); University of Arkansas (Other); Emory University (Other); St. Luke's Hospital and Health Network, Pennsylvania (Other); The Cleveland Clinic (Other); University of Tennessee (Other); TriHealth Inc. (Other); Tulane University (Other); Yale University (Other); Arrowhead Regional Medical Center (Other); Geisinger Clinic (Other); Miami Valley Hospital (Other)
Responsible Party: Principal Investigator, Alan Tita, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1U01HL119242-01 (NIH); U01HL119242-01 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-11-24 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: Pregnancy; Chronic hypertension
MeSH Terms: conditions — Hypertension | interventions — Labetalol; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-hypertensive therapy to goal <140/90 mmHg (Experimental): Labetalol or Nifedipine ER will be used as first-line to achieve goal; if necessary Nifedipine ER or Labetalol will be second-line antihypertensive. Rarely, other antihypertensive medications may also be used
  Interventions: Drug: Anti-hypertensive therapy
- No anti-hypertensive unless BP is severe (≥160/105 mmHg (Active Comparator): Antihypertensive therapy given only if BP becomes severe (defined as BP ≥160/105). The lowest dose of anti-hypertensive needed to keep blood pressure below this threshold will be given (1st-line - Labetalol or Nifedipine ER and 2nd-line - Labetalol or Nifedipine ER). Rarely other medications may be used
  Interventions: Other: No anti-hypertensive therapy (unless BP is severe)

INTERVENTIONS:
Drug: Anti-hypertensive therapy — 1st line anti-hypertensive (Labetalol or Nifedipine ER) started; escalate to maximum dose and a preferred 2nd line medication if needed (nifedipine ER or Labetalol)
  Other Names: Normodyne; Trandate; Procardia XL; Adalat
  Arms: Anti-hypertensive therapy to goal <140/90 mmHg
Other: No anti-hypertensive therapy (unless BP is severe) — Treatment will not be started if blood pressure remains <160/105; for blood pressure ≥160/105, treatment with labetalol or Nifedipine ER will be initiated and maintained at lowest dose needed to keep blood pressure under 160/105.
  Arms: No anti-hypertensive unless BP is severe (≥160/105 mmHg

SUMMARY:
The purpose of this study is to evaluate whether a blood pressure treatment strategy during pregnancy to achieve targets that are recommended for non-pregnant reproductive-age adults (<140/90 mmHg) compared ACOG- recommended standard during pregnancy (no treatment unless BP is severe) is effective and safe.

DETAILED DESCRIPTION:
During pregnancy, chronic hypertension (CHTN) is the most common major medical disorder encountered, occurring in 2-6%. The substantial negative effect of CHTN on pregnancy includes a consistent 3- to 5-fold increase in superimposed preeclampsia and adverse perinatal outcomes (fetal or neonatal death, preterm birth -PTB, poor fetal growth and placental abruption) and possibly a 5- to10-fold increase in maternal cardiovascular and other complications (death, cerebrovascular accident, pulmonary edema and acute renal failure). Mild CHTN (BP <160/110) contributes to a large proportion of these adverse outcomes. While antihypertensive treatment of CHTN is standard for the general population, it is uncertain whether treatment during pregnancy reduces maternal or fetal complications, and there are concerns that decreased arterial pressure may reduce fetal blood flow and cause poor fetal growth or small-for-gestational-age (SGA) infants. Some authorities, including the American College of Obstetricians and Gynecologists (ACOG) and American Society of Hypertension (ASH) recommend withholding antihypertensive therapy for mild CHTN, particularly if BP is <160/105-110 mmHg. The recommendation to withhold antihypertensive treatment in pregnancy conflicts with the broader public health goal to reduce BP in those with CHTN and there is no evidence that discontinuing therapy during the brief period of pregnancy affects maternal outcomes (other than reducing the severe hypertension). For over a decade, authorities have consistently called for well-designed and powered trials to delineate the benefits and risks of pharmacologic therapy for CHTN during pregnancy.

Therefore, our multicenter consortium proposes the Chronic Hypertension and Pregnancy (CHAP) Project, a large pragmatic randomized trial with a primary aim to evaluate the benefits and harms of pharmacologic treatment of mild CHTN in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Women with chronic hypertension in pregnancy with new or untreated chronic hypertension, blood pressure 140-159 systolic or 90-104 diastolic OR known chronic hypertension on monotherapy and taking any antihypertensive and blood pressure ≤159/104 (including those with blood pressure <140/90);
2. Singleton; and
3. viable pregnancy <23 weeks of gestation.

Exclusion Criteria:

1. Blood pressures prior to randomization ≥160 systolic or ≥105 diastolic (with or without treatment);
2. Severe hypertension including patients currently treated with >1 antihypertensive medication (more likely to have severe chronic hypertension);
3. Multi-fetal pregnancy;
4. Known secondary cause of chronic hypertension;
5. High-risk co-morbidities for which treatment may be indicated:

   * Diabetes mellitus diagnosed at age ≤10 years or duration of diagnosis ≥20 years
   * Diabetes mellitus complicated by end organ damage (retinopathy, nephropathy, heart disease, transplant)
   * Chronic kidney disease - including baseline proteinuria (>300mg/24-hr, protein/creatinine ratio ≥0.3, or persistent 1+ proteinuria*) or creatinine >1.2.

     *If a dipstick value at screening is more than trace, a clean catch or catheter urine should be obtained and re-tested by dipstick. If this shows trace or absence of protein, the patient is included. If it again shows 1+ protein, the patient is excluded until a 24-hr urine <300mg/24hr or p/c ratio is <0.3. If a p/c ratio is >0.3, the patient may be included if a 24-hour urine is < 300 mg.
   * Cardiac disorders: cardiomyopathy, angina, CAD
   * Prior stroke
   * Retinopathy
   * Sickle cell disease
6. Known major fetal anomaly;
7. Known fetal demise;
8. Suspected IUGR;
9. Membrane rupture or planned termination prior to randomization;
10. Plan to deliver outside the consortium centers (unless approved by the Clinical Coordinating Center) or unlikely to follow-up in the opinion of study staff or previous participation in this trial;
11. Contraindication to labetalol and nifedipine (e.g. know hypersensitivity);
12. Current substance abuse or addiction (cocaine, methamphetamine)
13. Participation in another trial without prior approval (CHAP participants will not be enrolled in other trials without prior approval by protocol committee)
14. Physician or provider refusal
15. Patient refusal *The minimum age varies by center

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2408 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tita, MD, PhD, Principal Investigator — University of Alabama at Birmingham - Clinical Coordinating Center; Gary Cutter, PhD, Principal Investigator — University of Alabama at Birmingham-Data Coordinating Center; Jeff Szychowski, PhD, Principal Investigator — University of Alabama at Birmingham-Data Coordinating Center
Locations (72):
- United States (72):
  - University of Alabama at Birmingham, Clinical Coordinating Center, Birmingham, Alabama
  - University of Alabama at Birmingham, Data Coordinating Center, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arrowhead Regional Medical Center, Colton, California
  - University of California, San Diego, San Diego, California
  - General Hospital of San Francisco, San Francisco, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Colorado, Boulder, Colorado
  - Denver Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern, Evanston, Illinois
  - Indiana University, Bloomington, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Lawrence, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Tulane, New Orleans, Louisiana
  - Ochsner Health System/Medical Center, New Orleans, Louisiana
  - Beaumont Hospital, Royal Oak, Michigan
  - University of Mississippi Medical College, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Peters University Hospital, New Brunswick, New Jersey
  - New Jersey Medical School, Newark, New Jersey
  - Virtua Medical Group, Sewell, New Jersey
  - New York Presbyterian Queens, Flushing, New York
  - Winthrop University Hospital, Mineola, New York
  - Columbia University, New York, New York
  - Weill Cornell, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke Regional Medical Center, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - WakeMed, Raleigh, North Carolina
  - TriHealth, Inc, Cincinnati, Ohio
  - Case Western/Metro Health, Cleveland, Ohio
  - Cleveland Clinic Fairview, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Cleveland Clinic-Hillcrest Hospital, Mayfield Heights, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Hospital/Health Network, Allentown, Pennsylvania
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburg/Magee Women's Center, Pittsburgh, Pennsylvania
  - Brown (WIHRI), Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - UT Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - UT Houston, Houston, Texas
  - McKay Dee Hospital, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Healthcare, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Gundersen Health System, La Crosse, Wisconsin
  - Unity Point Health-Meriter Hospital, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Research Institute, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Sanusi AA, Leach J, Boggess K, Dugoff L, Sibai B, Lawrence K, Hughes BL, Bell J, Aagaard K, Edwards RK, Gibson KS, Haas DM, Plante L, Metz TD, Casey B, Esplin S, Longo S, Hoffman MK, Saade GR, Hoppe KK, Foroutan J, Tuuli M, Owens MY, Simhan HN, Frey H, Rosen T, Palatnik A, Baker S, August P, Reddy UM, Su EJ, Krishna I, Nguyen NA, Norton ME, Skupski D, El-Sayed YY, Ogunyemi D, Galis ZS, Harper L, Ambalavanan N, Geller NL, Kuo HC, Sinkey RG, Librizzi R, Pereira L, Magann EF, Habli M, Williams S, Mari G, Pridjian G, McKenna DS, Parrish M, Eugene Chang, Osmundson S, Quinones J, Szychowski JM, Tita ATN. Pregnancy Outcomes of Nifedipine Compared With Labetalol for Oral Treatment of Mild Chronic Hypertension. Obstet Gynecol. 2024 Jul 1;144(1):126-134. doi: 10.1097/AOG.0000000000005613. Epub 2024 May 23. PMID 38949541
- [Derived] Moore MD, Kuo HC, Sinkey RG, Boggess K, Dugoff L, Sibai B, Lawrence K, Hughes BL, Bell J, Aagaard K, Edwards RK, Gibson KS, Haas DM, Plante L, Metz TD, Casey B, Esplin S, Longo S, Hoffman MK, Saade GR, Hoppe KK, Foroutan J, Tuuli M, Owens MY, Simhan HN, Frey HA, Rosen T, Palatnik A, Baker S, August P, Reddy UM, Kinzler W, Su EJ, Krishna I, Nguyen NA, Norton ME, Skupski D, El-Sayed YY, Ogunyemi D, Librizzi R, Pereira L, Magann EF, Habli M, Williams S, Mari G, Pridjian G, McKenna DS, Parrish M, Chang E, Osmundson S, Quinones JN, Leach J, Sanusi A, Galis ZS, Harper L, Ambalavanan N, Szychowski JM, Tita ATN. Mean Arterial Pressure and Neonatal Outcomes in Pregnancies Complicated by Mild Chronic Hypertension. Obstet Gynecol. 2024 Jul 1;144(1):101-108. doi: 10.1097/AOG.0000000000005611. Epub 2024 May 23. PMID 38781591
- [Derived] Bailey EJ, Tita ATN, Leach J, Boggess K, Dugoff L, Sibai B, Lawrence K, Hughes BL, Bell J, Aagaard K, Edwards RK, Gibson K, Haas DM, Plante L, Metz TD, Casey BM, Esplin S, Longo S, Hoffman M, Saade GR, Foroutan J, Tuuli MG, Owens MY, Simhan HN, Frey HA, Rosen T, Palatnik A, Baker S, August P, Reddy UM, Kinzler W, Su EJ, Krishna I, Nguyen N, Norton ME, Skupski D, El-Sayed YY, Ogunyemi D, Galis ZS, Harper L, Ambalavanan N, Oparil S, Kuo HC, Szychowski JM, Hoppe K. Perinatal Outcomes Associated With Management of Stage 1 Hypertension. Obstet Gynecol. 2023 Dec 1;142(6):1395-1404. doi: 10.1097/AOG.0000000000005410. Epub 2023 Sep 28. PMID 37769314
- [Derived] Goulding AN, Antoniewicz L, Leach JM, Boggess K, Dugoff L, Sibai B, Lawrence K, Hughes BL, Bell J, Edwards RK, Gibson K, Haas DM, Plante L, Metz TD, Casey B, Esplin S, Longo S, Hoffman M, Saade GR, Hoppe KK, Foroutan J, Tuuli M, Owens MY, Simhan HN, Frey H, Rosen T, Palatnik A, Baker S, Reddy UM, Kinzler W, Su E, Krishna I, Nguyen N, Norton ME, Skupski D, El-Sayed YY, Ogunyemi D, Harper LM, Ambalavanan N, Oparil S, Szychowski JM, Tita AT; Chronic Hypertension and Pregnancy Trial Consortium. Breastfeeding initiation and duration among people with mild chronic hypertension: a secondary analysis of the Chronic Hypertension and Pregnancy trial. Am J Obstet Gynecol MFM. 2023 Sep;5(9):101086. doi: 10.1016/j.ajogmf.2023.101086. Epub 2023 Jul 10. PMID 37437694
- [Derived] Tita AT, Szychowski JM, Boggess K, Dugoff L, Sibai B, Lawrence K, Hughes BL, Bell J, Aagaard K, Edwards RK, Gibson K, Haas DM, Plante L, Metz T, Casey B, Esplin S, Longo S, Hoffman M, Saade GR, Hoppe KK, Foroutan J, Tuuli M, Owens MY, Simhan HN, Frey H, Rosen T, Palatnik A, Baker S, August P, Reddy UM, Kinzler W, Su E, Krishna I, Nguyen N, Norton ME, Skupski D, El-Sayed YY, Ogunyemi D, Galis ZS, Harper L, Ambalavanan N, Geller NL, Oparil S, Cutter GR, Andrews WW; Chronic Hypertension and Pregnancy (CHAP) Trial Consortium. Treatment for Mild Chronic Hypertension during Pregnancy. N Engl J Med. 2022 May 12;386(19):1781-1792. doi: 10.1056/NEJMoa2201295. Epub 2022 Apr 2. PMID 35363951

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Started | 1208 | 1200
Completed | 1208 | 1200
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg | Total
Number analyzed (Participants) | 1208 | 1200 | 2408
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (5.6) | 32.3 (5.8) | 32.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1208 | 1200 | 2408
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or Ethnic Group: Non-Hispanic White | 347 | 326 | 673
  Race or Ethnic Group: Non-Hispanic Black | 574 | 570 | 1144
  Race or Ethnic Group: Hispanic | 238 | 250 | 488
  Race or Ethnic Group: Other | 49 | 54 | 103
Region of Enrollment [Number; unit: participants]
  United States | 1208 | 1200 | 2408
Insurance Type [Count of Participants; unit: Participants]
  Government-assisted or Medicaid | 673 | 656 | 1329
  Private | 459 | 463 | 922
  None | 60 | 65 | 125
  Missing data | 16 | 16 | 32
Type of CHTN [Count of Participants; unit: Participants]
  Newly diagnosed | 263 | 258 | 521
  Diagnosed and receiving medication | 677 | 681 | 1358
  Diagnosed and not receiving medication | 268 | 261 | 529
Blood Pressure - Systolic [Mean (Standard Deviation); unit: mmHg] | 134.3 (12.7) | 133.7 (12.4) | 134.0 (12.6)
Blood Pressure - Diastolic [Mean (Standard Deviation); unit: mmHg] | 83.9 (9.5) | 83.4 (9.6) | 83.7 (9.6)
Prior Pregnancy [Count of Participants; unit: Participants] | 1007 | 989 | 1996
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Data regarding body-mass index were missing for 19 in the active group and 22 in the control group.
  kg/m^2
    number analyzed (Participants) | 1189 | 1178 | 2367
    (all) | 37.7 (10.0) | 37.5 (9.6) | 37.6 (9.8)
Gestational Age less than 14 weeks [Count of Participants; unit: Participants] | 496 | 481 | 977
Diabetes Mellitus [Count of Participants; unit: Participants] | 191 | 189 | 380
Current Smoker [Count of Participants; unit: Participants] | 92 | 82 | 174
Aspirin Use [Count of Participants; unit: Participants] | 539 | 536 | 1075

OUTCOME MEASURES:

1. Primary Outcome: Composite Adverse Perinatal Outcome
Description: One or more severe outcomes including fetal death or neonatal death up to discharge or 90 days if prior; preeclampsia with severe features up to 2 weeks postpartum (Severe hypertension and proteinuria or hypertension and severe features per ACOG); placental abruption; or indicated PTB <35 weeks (not due to spontaneous preterm labor or membrane rupture).
Time Frame: Up to 2 weeks postpartum for preeclampsia or 90 days for neonatal death
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1170 | 1155
Participants
  Composite Primary Outcome | 353 | 427
  Preeclampsia with Severe Features | 272 | 336
  Indicated Preterm Birth <35 weeks | 143 | 193
  Placental Abruption | 20 | 22
  Fetal or Neonatal Death <28 days | 41 | 50
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; p < 0.001, Chi-squared; Risk Ratio (RR) = .82, 95% CI 2-sided [.73 to .92]
Statistical Analysis 2: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .80, 95% CI 2-sided [.70 to .90]
Statistical Analysis 3: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .73, 95% CI 2-sided [.60 to .89]
Statistical Analysis 4: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .90, 95% CI 2-sided [.49 to 1.64]
Statistical Analysis 5: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .81, 95% CI 2-sided [.54 to 1.21]

2. Primary Outcome: Small for Gestational Age (Safety)
Description: Birth weight less than 10th percentile for gestational age at birth according to accepted national standard
Time Frame: Until delivery
Population: Analysis is restricted to 2270 (1146 in the Treatment Group and 1124 in the Standard Group) who were delivered and who had complete assessments during delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1146 | 1124
Participants | 128 | 117
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; p = 0.56, Chi-squared; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.85 to 1.36]

3. Secondary Outcome: Composite of Maternal Death or Severe Cardiovascular Morbidity
Description: One or more of maternal death, new heart failure, stroke, encephalopathy, angina, myocardial infarction or ischemia, pulmonary edema, ICU admission/intubation, or renal failure
Time Frame: Up to 6 weeks (4-12 weeks) after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 25 | 33
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .75, 95% CI 2-sided [.45 to 1.26]

4. Secondary Outcome: Severe Maternal Hypertension + Components of the Primary Composite Endpoint
Description: Persistent severe hypertension with or without proteinuria + the primary composite
Time Frame: Up to 2 weeks postpartum or 90 days for neonatal death
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 529 | 631
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.77 to 0.91]

5. Secondary Outcome: Preterm Birth and Indicated Preterm Birth (<37 Weeks)
Description: Preterm birth and Indicated preterm birth (<37 weeks) includes any preterm birth less than 37 weeks
Time Frame: Until delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 332 | 377
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .87, 95% CI 2-sided [.77 to .99]

6. Secondary Outcome: Composite of Severe Neonatal Morbidities
Description: One or more of Bronchopulmonary dysplasia (BPD), Retinopathy of prematurity (ROP), Necrotizing enterocolitis (NEC), Intraventricular hemorrhage (VH) grade III/IV
Time Frame: Up to 90 days post delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 24 | 31
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .77, 95% CI 2-sided [.45 to 1.3]

7. Secondary Outcome: Adherence to Treatment After Delivery
Description: Counts with high adherence to antihypertensive therapy after delivery for those prescribed medications.
Time Frame: 6 weeks (4-12 weeks) after delivery
Population: Analysis is restricted to 706 in Treatment Group and 479 in Standard Group who had complete antihypertensive therapy assessments at the follow-up study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 706 | 479
Participants | 436 | 275
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = 1.08, 95% CI 2-sided [.98 to 1.18]

8. Other Pre Specified Outcome: Superimposed Preeclampsia
Description: Mild or severe, including eclampsia
Time Frame: Up to 2 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 295 | 373
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .79, 95% CI 2-sided [.69 to .89]

9. Other Pre Specified Outcome: Superimposed Gestational Hypertension
Description: Persistent worsening hypertension above baseline without pree or proteinuria occurring after 20 weeks gestation
Time Frame: Enrollment (between 6 and 18 weeks gestation) to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 132 | 156
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.68 to 1.04]

10. Other Pre Specified Outcome: Severe Hypertension
Description: Blood pressure ≥160/110
Time Frame: Up to 6 weeks (4-12 weeks) after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 436 | 531
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .82, 95% CI 2-sided [.74 to .90]

11. Other Pre Specified Outcome: Cesarean Delivery
Description: Cesarean delivery
Time Frame: Until delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 592 | 582
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [.93 to 1.10]

12. Other Pre Specified Outcome: Blood Transfusion
Description: During pregnancy or postpartum
Time Frame: Up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 46 | 53
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .86, 95% CI 2-sided [.59 to 1.27]

13. Other Pre Specified Outcome: NICU Admission
Description: Any NICU admission
Time Frame: Up to 6 weeks (4-12 weeks) after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 368 | 402
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .91, 95% CI 2-sided [.81 to 1.02]

14. Other Pre Specified Outcome: Low Birth Weight
Description: Birth weight <2500g
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 232 | 277
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .83, 95% CI 2-sided [.71 to .97]

15. Other Pre Specified Outcome: Ponderal Index
Description: Mean ponderal index, mass/height^3 at birth
Time Frame: At birth
Population: data incomplete for 71 in the Treated Group and 83 in the Standard Group
Measure: Mean (Standard Deviation); unit: g/cm^3
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1137 | 1117
g/cm^3 | 2.9 (3.7) | 2.7 (2.8)
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Mean Difference (Final Values) = .16, 95% CI 2-sided [-0.11 to 0.43]

16. Other Pre Specified Outcome: Head Circumference
Description: Mean head circumference
Time Frame: At birth
Population: data incomplete for 84 in the Treated Group and 97 in the Standard Group
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1124 | 1103
cm | 33.3 (3.0) | 33.0 (3.0)
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [0.05 to 0.56]

17. Other Pre Specified Outcome: Placental Weight
Description: Mean placental weight
Time Frame: At delivery
Population: data incomplete for 549 in the Treated Group and 562 in the Standard Group
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 659 | 638
g | 466.3 (177.6) | 464.6 (175.6)
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-17.6 to 20.9]

18. Other Pre Specified Outcome: Hypoglycemia
Description: Prevalence of hypoglycemia
Time Frame: From delivery to hospital discharge (2 - 3 days after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 191 | 195
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .97, 95% CI 2-sided [.81 to 1.17]

19. Other Pre Specified Outcome: Bradycardia
Description: Prevalence of bradycardia
Time Frame: From delivery to hospital discharge (2 - 3 days after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 31 | 35
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .88, 95% CI 2-sided [.55 to 1.42]

20. Other Pre Specified Outcome: Hypotension
Description: Incidence (%) with hypotension
Time Frame: From delivery to hospital discharge (2 - 3 days after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 7 | 16
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .43, 95% CI 2-sided [.18 to 1.05]

21. Other Pre Specified Outcome: Respiratory Distress Syndrome (RDS)
Description: Incidence (%) with respiratory distress syndrome (RDS)
Time Frame: From delivery to hospital discharge (2 - 3 days after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 149 | 171
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .87, 95% CI 2-sided [.71 to 1.06]

22. Other Pre Specified Outcome: Bronchopulmonary Dysplasia (BPD)
Description: Incidence (%) with bronchopulmonary dysplasia (BPD)
Time Frame: Up to 3 months after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 8 | 14
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .57, 95% CI 2-sided [.24 to 1.35]

23. Other Pre Specified Outcome: Intubation/Ventilation
Description: Incidence (%) with resuscitation including oxygen, intubation, chest compression/CPR, or CPAP
Time Frame: From delivery to hospital discharge (2 - 3 days after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 298 | 303
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .98, 95% CI 2-sided [.85 to 1.12]

24. Other Pre Specified Outcome: Intraventricular Hemorrhage (IVH)
Description: Incidence (%) with any IVH and with IVH Grades III and IV
Time Frame: From delivery to hospital discharge (2 - 3 days after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 11 | 17
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.30 to 1.37]

25. Other Pre Specified Outcome: Necrotizing Enterocolitis (NEC)
Description: Incidence (%) with necrotizing enterocolitis (NEC)
Time Frame: Up to 3 months after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 2 | 2
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .99, 95% CI 2-sided [.14 to 7.06]

26. Other Pre Specified Outcome: Hyperbilirubinemia
Description: Incidence (%) with hyperbilirubinemia
Time Frame: From delivery to hospital discharge (2 - 3 days after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 266 | 283
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .93, 95% CI 2-sided [.81 to 1.08]

27. Other Pre Specified Outcome: 5-min Apgar Score
Description: Incidence (%) with Apgar score <7 (range 0-10 with lower scores indicating worse outcome)
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 68 | 80
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .84, 95% CI 2-sided [0.62 to 1.16]

28. Other Pre Specified Outcome: Sepsis
Description: Incidence (%) with proven sepsis
Time Frame: From delivery to hospital discharge (2 - 3 days after delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 21 | 34
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = .61, 95% CI 2-sided [.36 to 1.05]

29. Other Pre Specified Outcome: Unscheduled Prenatal Clinic or ER Visits
Description: Number of unscheduled clinic or ER visits before and after delivery
Time Frame: Up to 3 months after delivery
Measure: Mean (Standard Deviation); unit: number of encounters
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
number of encounters | 1.1 (1.6) | 1.2 (1.6)
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.2 to 0.03]

30. Other Pre Specified Outcome: Hospitalizations
Description: Number of hospitalizations before or after delivery
Time Frame: Up to 3 months postpartum
Measure: Mean (Standard Deviation); unit: number of encounters
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
number of encounters | 0.3 (0.7) | 0.3 (0.8)
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.1 to 0.1]

31. Other Pre Specified Outcome: Postpartum Unscheduled or ER Visits
Description: Number of postpartum unscheduled or ER visits
Time Frame: Up to 3 months after delivery
Measure: Mean (Standard Deviation); unit: number of encounters
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
number of encounters | 0.3 (0.8) | 0.4 (0.8)
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.12 to 0.002]

32. Other Pre Specified Outcome: Postpartum Hospitalizations
Description: Number of postpartum hospitalizations
Time Frame: Up to 3 months after delivery
Measure: Mean (Standard Deviation); unit: number of encounters
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
number of encounters | 0.15 (0.44) | 0.14 (0.37)
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.02 to 0.04]

33. Other Pre Specified Outcome: Neonatal Hospital Stay of 3 or More Days
Description: Frequency of neonatal hospital stays lasting at least 3 days
Time Frame: after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
Number analyzed (Participants) | 1208 | 1200
Participants | 590 | 592
Statistical Analysis 1: Comparison: Anti-hypertensive Therapy to Goal <140/90 mmHg vs No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.90 to 1.06]

ADVERSE EVENTS:
Time Frame: Adverse event data collected up to 2 week postpartum visit.
Arm/Group | Anti-hypertensive Therapy to Goal <140/90 mmHg | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg
All-Cause Mortality (participants affected / at risk) | 42/1208 | 52/1200
Serious Adverse Events (participants affected / at risk) | 113/1208 | 126/1200
Other Adverse Events (participants affected / at risk) | 0/1208 | 0/1200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-hypertensive Therapy to Goal <140/90 mmHg (N=1208) | No Anti-hypertensive Unless BP is Severe (≥160/105 mmHg (N=1200)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Foetal anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 36 (36) | 42 (42)
Foetal Growth Restriction (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 24 (24)
Death Neonatal (General disorders) | 5 (5) | 8 (8)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 19 (19)
Maternal Death (General disorders) | 1 (1) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Congenital Pneumonia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gestational Hypertension (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary Oedema (Reproductive system and breast disorders) | 4 (4) | 5 (5)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 4 (4)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Gravitational Oedema (General disorders) | 0 (0) | 1 (1)
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HELLP Syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hyperbilirubinaemia Neonatal (Hepatobiliary disorders) | 3 (3) | 0 (0)
Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Bronchopulmonary Dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0)
Cleft Lip and Palate (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital Genitourinary Abnormality (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital Diaphragmatic Hernia (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Diaphragmatic Aplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Holoprosencephaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Neonatal Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Neonatal Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oesophageal Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Placenta Accreta (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postpartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Preterm Premature Rupture of Membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Shoulder Dystocia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Trisomy 21 (Congenital, familial and genetic disorders) | 2 (2) | 3 (3)
Ventricular Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Trisomy 18 (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Multiple Cardiac Defects (Congenital, familial and genetic disorders) | 2 (2) | 4 (4)
Renal Aplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 3 (3) | 1 (1)
Microcephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Dandy-Walker syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypoplastic Left Heart Syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Kidney Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Anomalous Pulmonary Venous Connection (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Chondrodystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage Neonatal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Shortened Cervix (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Renal Tubular Necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Purulent Discharge (Infections and infestations) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Foetal Chromosome Abnormality (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Uterine rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure abnormal (Investigations) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Fetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Poor weight gain neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abdominal operation (Surgical and medical procedures) | 2 (2) | 0 (0)
General Event (General disorders) | 12 (12) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT02299414/Prot_SAP_000.pdf